CLINICAL TRIAL: NCT02353559
Title: Emotion And Symptom-focused Engagement (EASE): A Randomized Pilot Trial of an Intervention for Individuals With Acute Leukemia
Brief Title: Emotion And Symptom-focused Engagement (EASE): An Intervention for Individuals With Acute Leukemia
Acronym: EASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-6631
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Acute Leukemia
Keywords: acute leukemia; traumatic stress; quality of life; symptom burden; psychosocial oncology; palliative care; intervention; hematological malignancies; supportive care
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EASE (Experimental): Patients assigned to the intervention arm will receive 8 - 12 psychotherapy sessions lasting 30 - 60 minutes each, delivered by a trained therapist at our center. Patients will receive specialized symptom control from a nurse/physician team in our Palliative Care Service, when indicated by routine symptom screening.
  Interventions: Behavioral: EASE
- Usual Care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: EASE — EASE includes psychotherapeutic (EASE-psy) and physical symptom control (EASE-phys) components.
  Arms: EASE

SUMMARY:
The purpose of this study is to test the feasibility of an individual psychological and physical symptom intervention, called Emotion And Symptom-focused Engagement (EASE), to reduce traumatic stress and physical symptom burden in individuals newly diagnosed with acute leukemia.

DETAILED DESCRIPTION:
This study involves the pilot-testing of a newly developed, brief manualized individual psychotherapy and physical symptom control intervention, called Emotion And Symptom-focused Engagement (EASE), to reduce traumatic stress and physical symptom burden in individuals newly diagnosed with acute leukemia. The purpose of this study is to conduct a two-arm randomized pilot trial (RPT) to test the feasibility, acceptability, and preliminary efficacy of EASE against usual care (UC) for the reduction of traumatic stress and physical symptom burden in patients with acute leukemia. Usual care for individuals with acute leukemia treated at the Princess Margaret Cancer Centre includes referral for non-standardized, and primarily instrumental, psychosocial care and palliative care service as needed.

The design will be an unblinded RPT consisting of two conditions (EASE and UC), with a baseline assessment and follow-ups at 4, 8, and 12 weeks. The trial will take place at the Princess Margaret Cancer Centre, University Health Network; a comprehensive cancer center in Toronto, Canada. Participants will be newly diagnosed with acute leukemia, within one month of diagnosis and/or admission to hospital for treatment with curative intent.

ELIGIBILITY:
Inclusion Criteria:

* new or relapsed diagnosis of acute leukemia (an amendment to allow recruitment of relapsed patients was approved on 24-Sep-2015, although no relapsed patients were ultimately recruited)
* will be receiving induction chemotherapy with curative intent and within 1 month of diagnosis and/or admission to hospital at the Princess Margaret Cancer Centre
* age ≥ 18 years
* fluency in English
* no cognitive impairment indicated in the medical record, communicated by the hematology clinical team, or determined by research staff at recruitment.

Exclusion Criteria:

* inability to pass the cognitive screening test (Short Orientation-Memory Concentration Test [SOMC] score <20)
* actively receiving psychological/psychiatric counseling or palliative care services from the Department of Psychosocial Oncology and Palliative Care (POPC), now called the Department of Supportive Care, at the Princess Margaret Cancer Centre at the time of recruitment to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Stanford Acute Stress Reaction Questionnaire (SASRQ) | 12 weeks
  A 30-item reliable and valid self-report measure of traumatic stress symptoms.

SECONDARY OUTCOMES:
Functional Assessment of Chronic Illness Therapy-Spiritual Well-Being Scale (FACIT-Sp) | 12 weeks
  A 40-item reliable and valid self-report measure of overall quality of life, including 12 items that assess spiritual well-being, spiritual meaning and peace, and faith.
Beck Depression Inventory-II (BDI-II) | 12 weeks
  A 21-item reliable and valid self-report measure of the intensity of depressive symptoms, consistent with the DSM-V criteria for major depressive disorder.
Brief Pain Inventory short form (BPI-sf) | 12 weeks
  A 9-item reliable and valid self-report measure that assesses pain severity and the impact of pain on daily functioning.
Memorial Symptom Assessment Scale (MSAS) | 12 weeks
  A 32-item reliable and valid self-report inventory assessing the presence and severity of 26 common physical symptoms and 6 psychological symptoms of cancer. The scale has been adapted to reduce burden. A shortened version that omits frequency of symptoms and treatment, and satisfaction with treatment for each symptom was used.
Brief Experiences in Close Relationships Scale (ECR-M16) | 12 weeks
  A 16-item reliable and valid self-report measure of attachment security.
FAMCARE-P16 | 12 weeks
  A 16-item reliable and valid self-report measure of patient satisfaction with healthcare providers.
Clinical Evaluation Questionnaire (CEQ) | 12 weeks
  A 7-item measure developed for this study to evaluate the extent to which patients felt emotionally supported by the clinical services provided.
Edmonton Symptom Assessment System - Acute Leukemia (ESAS-AL) | 24 hours
  A 14-item symptom severity assessment measure adapted for patients with acute leukemia to include prevalent and treatable symptoms in this population: mouth sores, diarrhea, itching, constipation, and insomnia. ESAS-AL was used as a screening tool as part of the clinical intervention, and was added as an outcome later in the trial (13-Apr-2016).

CONTACTS AND LOCATIONS:
Overall Officials: Gary Rodin, MD FRCPC, Principal Investigator — University Health Network, Toronto; Camilla Zimmermann, MD PhD FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Rodin G, Yuen D, Mischitelle A, Minden MD, Brandwein J, Schimmer A, Marmar C, Gagliese L, Lo C, Rydall A, Zimmermann C. Traumatic stress in acute leukemia. Psychooncology. 2013 Feb;22(2):299-307. doi: 10.1002/pon.2092. Epub 2011 Nov 13. PMID 22081505
- [Background] Zimmermann C, Swami N, Krzyzanowska M, Hannon B, Leighl N, Oza A, Moore M, Rydall A, Rodin G, Tannock I, Donner A, Lo C. Early palliative care for patients with advanced cancer: a cluster-randomised controlled trial. Lancet. 2014 May 17;383(9930):1721-30. doi: 10.1016/S0140-6736(13)62416-2. Epub 2014 Feb 19. PMID 24559581
- [Background] Zimmermann C, Yuen D, Mischitelle A, Minden MD, Brandwein JM, Schimmer A, Gagliese L, Lo C, Rydall A, Rodin G. Symptom burden and supportive care in patients with acute leukemia. Leuk Res. 2013 Jul;37(7):731-6. doi: 10.1016/j.leukres.2013.02.009. Epub 2013 Mar 11. PMID 23490030
- [Background] Nissim R, Zimmermann C, Minden M, Rydall A, Yuen D, Mischitelle A, Gagliese L, Schimmer A, Rodin G. Abducted by the illness: a qualitative study of traumatic stress in individuals with acute leukemia. Leuk Res. 2013 May;37(5):496-502. doi: 10.1016/j.leukres.2012.12.007. Epub 2013 Jan 24. PMID 23352641
- [Background] Nissim R, Rodin G, Schimmer A, Minden M, Rydall A, Yuen D, Mischitelle A, Fitzgerald P, Lo C, Gagliese L, Zimmermann C. Finding new bearings: a qualitative study on the transition from inpatient to ambulatory care of patients with acute myeloid leukemia. Support Care Cancer. 2014 Sep;22(9):2435-43. doi: 10.1007/s00520-014-2230-3. Epub 2014 Apr 5. PMID 24705856
- [Background] Zimmermann C, Seccareccia D, Clarke A, Warr D, Rodin G. Bringing palliative care to a Canadian cancer center: the palliative care program at Princess Margaret Hospital. Support Care Cancer. 2006 Oct;14(10):982-7. doi: 10.1007/s00520-006-0093-y. Epub 2006 Jun 27. PMID 16802127
- [Background] Rodin G, Deckert A, Tong E, Le LW, Rydall A, Schimmer A, Marmar CR, Lo C, Zimmermann C. Traumatic stress in patients with acute leukemia: A prospective cohort study. Psychooncology. 2018 Feb;27(2):515-523. doi: 10.1002/pon.4488. Epub 2017 Aug 10. PMID 28665521
- [Background] Shaulov A, Rodin G, Popovic G, Caraiscos VB, Le LW, Rydall A, Schimmer AD, Zimmermann C. Pain in patients with newly diagnosed or relapsed acute leukemia. Support Care Cancer. 2019 Aug;27(8):2789-2797. doi: 10.1007/s00520-018-4583-5. Epub 2018 Dec 8. PMID 30535882
- [Result] Rodin G, Malfitano C, Rydall A, Schimmer A, Marmar CM, Mah K, Lo C, Nissim R, Zimmermann C. Emotion And Symptom-focused Engagement (EASE): a randomized phase II trial of an integrated psychological and palliative care intervention for patients with acute leukemia. Support Care Cancer. 2020 Jan;28(1):163-176. doi: 10.1007/s00520-019-04723-2. Epub 2019 Apr 17. PMID 31001692